CLINICAL TRIAL: NCT01063296
Title: Effects of Chemotherapy on Circulating Tumor Cells and Recurrences in IB-IIA Cervical Cancer Patients With Intermediate Risk Factors After Radical Surgery
Brief Title: Effects of Chemotherapy on Circulating Tumor Cells and Recurrences in Cervical Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Ding Ma, Cancer Biology Research Center of Tongji Hospital
Other Study IDs: GM2010-02
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-01

CONDITIONS: Cervical Cancer
Keywords: cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sampling of peripheral blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cervical cancer is a major health problem for Chinese women. It is estimated that nearly 100,000 new cervical cancer cases occur in China every year, which accounts for about 20 percent of global new cases. Surgery and radiotherapy are two major radical treatment methods for IB-IIB cervical cancer. Unlike the United States and some other countries, most of operable women with IB-IIB cervical cancer received radical surgery other than radiotherapy in China. Patients with recurrence risk factors (lymph node metastasis, deep stromal invasion, positive lymphatic vascular space, et al. ) also received adjuvant therapy after surgery, such as radiotherapy or chemoradiotherapy that are recommended in the NCCN guidelines. However, in China a substantial part of patients especially those admitted to tertiary hospitals received several courses of chemotherapy instead of radiotherapy if they had recurrence risk factors .

In our previous study, we found that patients with intermediate risk factors (deep stromal invasion, positive lymphatic vascular space, bulky tumor>4cm) had better disease-free survival and recurrence-free survival when they received chemotherapy compared with radiotherapy. The objective in this study is to investigate whether the advantage of postoperative chemotherapy is a result of circulating tumor cells (CTC) in some of the patients with intermediate risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed Ib~IIa （FIGO）cervical carcinoma without previous treatments
* Age between 18-70
* With the presence of these three pathological risk factors after radical surgery:(1) positive lymphatic vascular space,(2)outer one-third invasion of the cervical stroma, (3) bulky tumor≥4cm
* At least 3 months of disease-free survival

Exclusion Criteria:

* The presence of other uncontrolled life-threatening disease (Suffering from myocardial infarction or stroke, or unstable angina, decompensated heart failure, or a history of deep vein thrombosis)
* Receiving other anti-cancer therapy, such as traditional Chinese drug
* Don't be able to finish the whole treatment(chemotherapy or radiotherapy)
* liver dysfunction (ALT、AST>2.5×ULN)
* renal dysfunction (Creatinine>1.5×ULN)
* WBC<4,000/mm3 or PLT<100,000/mm3
* Received preoperative radiotherapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed Ib~IIa cervical carcinoma without previous treatments
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence rate of CTCs, distant metastasis-free survival, disease-free survival, metastatic sites | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ma Ding, M.D., Study Director — Tongji Hospital of HUST
Locations (1):
- Tongji Hospital of HUST, Wuhan, Hubei, China